CLINICAL TRIAL: NCT04921917
Title: The Effect of Exercise on Patient Outcomes During Treatment of Soft Tissue Sarcoma With Neoadjuvant Radiation Therapy and Surgical Resection
Brief Title: Exercise and Soft Tissue Sarcoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00093033
Record Dates: First submitted 2021-05-18; First posted 2021-06-10 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Soft Tissue Sarcoma
Keywords: exercise; soft tissue sarcoma; STS
MeSH Terms: conditions — Sarcoma; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This study is partially blinded. The wound surveyor and statistician(s) will be blinded to the treatment groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard of care: neoadjuvant radiation therapy (NRT).
- Neoadjuvant Exercise Regimen (Experimental): Subjects will receive conventional NRT in conjunction with a prescribed exercise regimen during the usual 10-week duration of NRT treatment prior to tumor resection.
  Interventions: Other: neoadjuvant exercise therapy

INTERVENTIONS:
Other: neoadjuvant exercise therapy — brief exercise regimen completed immediately prior to neoadjuvant radiation therapy. Rubber bands will be used for the exercise training of patients with lower extremity tumors while an electronic hand-held dynamometer will be used for the exercise training for patients with upper extremity tumors.
  Arms: Neoadjuvant Exercise Regimen

SUMMARY:
The purpose of this study is to evaluate the effect of a neoadjuvant (i.e. pre-treatment) exercise regimen on extremity function and postoperative wound healing. The study group will include patients with a primary diagnosis of soft tissue sarcoma undergoing treatment with neoadjuvant radiation therapy and surgical resection. Patients with upper or lower extremity sarcomas will be considered for enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females within the ages of 18-85
2. Diagnosis of soft tissue sarcoma that has been histologically confirmed by an approved reference pathologist
3. Sarcoma of the upper or lower extremity location
4. Treatment plan that includes neo-adjuvant radiation therapy followed by surgical resection
5. Expected primary wound closure performed at the time at surgery
6. Any disease stage
7. Any tumor grade
8. Any histologic subtype
9. First or recurrent presentations
10. No vascular invasion or resection/repair/reconstruction that results in decreased perfusion of the extremity
11. No history of radiation therapy to the tumor and/or surgical area prior to the current treatment being studied
12. Must be able to comply with follow up visits
13. Must be able to provide own consent

Exclusion Criteria:

1. Patients under the age of 18, or over the age of 85
2. Treatment plan that does not include neo-adjuvant radiation and surgical excision
3. Sarcoma location other than the upper or lower extremity
4. History of radiation therapy to the tumor and/or surgical area prior to the current treatment being studied
5. High dose steroid therapy (defined as >5mg prednisone, or equivalent, with the last 30 days)
6. Active treatment with chemotherapy within the last 30 days
7. Inability of the patient to provide informed consent (i.e. dementia, cognitive impairment, non-English speakers)
8. Plan for post-operative radiation therapy
9. Underlying severe cardiopulmonary disease
10. Prior surgery, other than a biopsy, at the site of disease
11. Tumors that are ulcerative or fungating through the dermis at the time of presentation
12. Vascular invasion or resection/repair/reconstruction that results in decreased perfusion of the extremity
13. Vascular disease resulting in clinically apparent compromise in blood flow to the treatment extremity (i.e. peripheral vascular disease with diminished pulses, venous insufficiency with clinical evidence of vascular congestion)
14. Actively uncontrolled diabetes mellitus (documentation of history of Diabetes with A1c>8)
15. Active deep vein thrombosis in the treatment extremity
16. Inability to comply with follow up visits
17. Pregnant females (women of childbearing potential must have a negative serum pregnancy test prior to enrollment)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with a wound complication after surgery as measured by wound complication form | Up to 24 weeks post-op
  The wound complication form is a team developed form that asks about different complications that can arise after surgery. These complications include delayed wound healing, surgical site or periprosthetic infection, re-operation, and other invasive procedures necessitated by wound complications.

SECONDARY OUTCOMES:
Percent necrosis of tumor | During surgery
  Percent necrosis at the time of tumor resection
Number of inflammatory serum markers | First day of NRT
  Number of inflammatory serum markers as assessed by CRP, Complete Blood Count, and ESR.
Number of inflammatory serum markers | Halfway through NRT (up to 5 weeks of NRT)
  Number of inflammatory serum markers as assessed by CRP, Complete Blood Count, and ESR.
Number of inflammatory serum markers | Last day of NRT (up to 10 weeks of NRT)
  Number of inflammatory serum markers as assessed by CRP, Complete Blood Count, and ESR.
Tissue Perfusion | 6-week post-op
  Tissue Perfusion using the Near Infra-Red (NIRS) system
The Musculoskeletal Tumor Society (MSTS) score | At enrollment.
  The Musculoskeletal Tumor Society (MSTS) score of extremity function. The total score ranges from 0 to 30, with higher scores indicating better function.
The Musculoskeletal Tumor Society (MSTS) score | 2 weeks or less prior to surgery
  The Musculoskeletal Tumor Society (MSTS) score of extremity function. The total score ranges from 0 to 30, with higher scores indicating better function.
The Musculoskeletal Tumor Society (MSTS) score | 6-week post-op
  The Musculoskeletal Tumor Society (MSTS) score of extremity function. The total score ranges from 0 to 30, with higher scores indicating better function.
Edmonton Symptom Assessment System (ESAS) - Sarcoma Modified (SM) quality of life questionnaire | At enrollment
  The Edmonton Symptom Assessment System - Sarcoma Modified (ESAS-SM) questionnaire on quality of life. The total score ranges from 0 to 110, with lower scores indicating better quality of life.
Edmonton Symptom Assessment System (ESAS) - Sarcoma Modified (SM) quality of life questionnaire | 2 weeks or less prior to surgery
  The Edmonton Symptom Assessment System - Sarcoma Modified (ESAS-SM) questionnaire on quality of life. The total score ranges from 0 to 110, with lower scores indicating better quality of life.
Edmonton Symptom Assessment System (ESAS) - Sarcoma Modified (SM) quality of life questionnaire | 6-week post-op
  The Edmonton Symptom Assessment System - Sarcoma Modified (ESAS-SM) questionnaire on quality of life. The total score ranges from 0 to 110, with lower scores indicating better quality of life.
Surgical Wound Assessment Form | Up to 24 weeks post-op
  Wound assessment and healing tracker tool created by the study team. The total score ranges from 13 to 65, with lower scores indicating better wound healing.

CONTACTS AND LOCATIONS:
Overall Officials: William Eward, DVM, MD, Principal Investigator — Duke Orthopedic Oncology
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No